CLINICAL TRIAL: NCT06053502
Title: The Filtering Facepiece Respirator Increases Inspiratory Time, But Does Not Change the Involvement of Breathing Compartments
Brief Title: Respirator and Breathing Compartments
Acronym: Breathing
Status: Completed | Type: Observational
Sponsor: University of South Bohemia (Other)
Responsible Party: Sponsor
Other Study IDs: KPTVSPFJUAugust2023
Record Dates: First submitted 2023-08-28; First posted 2023-09-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Face Mask Squeeze; Respiratory Complication
Keywords: optoelectronic plethysmography; breathing compartments; N95; graded exercise test

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Masked condition: Participants who underwent the graded exercise test with the respirator.
  Interventions: Other: filtering facepiece respirator
- Unmasked condition: Participants who underwent the graded exercise test without the respirator.

INTERVENTIONS:
Other: filtering facepiece respirator — Graded exercise test with filtering facepiece respirator
  Groups: Masked condition

SUMMARY:
The purpose of this study was to compare breathing pattern and involvement of individual breathing compartments (IBC) with and without filtering facepiece respirator (FFR) during rest and exercise.

DETAILED DESCRIPTION:
The study involved 21 students majoring in physical education and sports. All subjects were physically active, engaging in approximately 260 minutes of physical activity per week, and they possessed a high level of fitness. Inclusion criteria required participants to be free from injury, capable of providing written consent, and within the age range of 19 to 26 years. Exclusion criteria included individuals who smoked or had chronic pulmonary or cardiac diseases. This research received approval from the Ethics Committee at the Faculty of Education, University of South Bohemia, Reference Number: 002/2018. All procedures conducted within the study adhered to the ethical standards outlined by the Institutional Research Committee and the principles of the Helsinki Declaration.

Protocol:

Participants were instructed to visit the laboratory on two occasions to complete two separate tests during each session, specifically the Opto-electronic plethysmography (OEP) test during resting in a standing position and the OEP test during a Graded Exercise Test (GXT). The time interval between the testing days was three days. Participants were randomly assigned to two groups using randomizer.org. The first group performed three tests while wearing a Face-Fit Respirator (FFR), while the second group performed the tests without the mask. During the second visit, participants switched to the opposite condition. The N95 respirator was employed in this study as the gold standard for protection against aerosol transmission, particularly during the COVID-19 pandemic. A new mask was used for each test. In the Standing Test (STD), participants were instructed to maintain a stationary standing position and engage in spontaneous, quiet breathing without speaking or altering their posture while OEP data was collected. The first two minutes were designated as an adaptation period, followed by data collection for an additional three minutes. In the context of the Graded Exercise Test (GXT), OEP data was collected during the final minute of each three-minute stage.

Opto-Electronic Plethysmography:

The analysis of breathing patterns and volumes of chest wall compartments was conducted using opto-electronic plethysmography (BTS Bioengineering, Milan, Italy). This device comprises eight cameras, with five positioned anteriorly and three posteriorly relative to the participant. Additionally, 89 reflective markers were affixed to the participant's chest, abdomen, and back to track movements of the trunk. This technique has previously demonstrated validity in both resting and maximal exercise conditions.

The contributions of each breathing compartment (VRCp - pulmonary rib cage, VRCa - abdominal rib cage, VAb - abdomen) were determined by calculating the difference between end-inspiratory and end-expiratory volumes. The specific methodology for calculating chest wall kinematics using OEP has been detailed in prior research.

Graded Exercise Tests:

To complete this study, participants were required to undergo two maximal graded exercise tests (GXT) on separate days, one with the use of a Face-Fit Respirator (FFR) and one without. After three minutes of warm-up walking (2.7 km/h, 10% incline), participants performed the Bruce Protocol until exhaustion. The Bruce Protocol was conducted on a treadmill (Lode Valiant 2 Sport, Lode B.V., Groningen, Netherlands). All tests were conducted at the same time of day to mitigate the influence of circadian rhythms. Immediately following the completion of the test, participants provided ratings on the Modified Borg Dyspnea Scale, which ranges from 0 to 10, to assess breathlessness.

ELIGIBILITY:
Inclusion Criteria:

* physically active (~260 min/week) possessing high fitness level,
* free from injury,
* able to give full written consent,
* meet age criteria 19-26 years.

Exclusion Criteria:

* smokers,
* chronic pulmonary disease,
* cardiac disease.

Ages: 19 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students of physical education and sport
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-08-26 (Actual)

PRIMARY OUTCOMES:
Inspiratory time | up to 12 weeks
  Inspiratory time in every phase of the GXT will be presented as a mean and standard deviation, along with the mean difference and a 95% confidence interval of the difference. Inspiratory time will be measured using opto-electronic plethysmography, with units in [s], and the outcomes will be compared using a repeated-measures ANOVA with intra-subject comparisons.
Expiratory time | up to 12 weeks
  Expiratory time in every phase of the GXT will be presented as a mean and standard deviation, along with the mean difference and a 95% confidence interval of the difference. Expiratory time will be measured using opto-electronic plethysmography, with units in [s], and the outcomes will be compared using a repeated-measures ANOVA with intra-subject comparisons.
Chest wall compartments | up to 12 weeks
  The individual contribution of chest wall compartments in every phase of the GXT will be presented as a mean and standard deviation, along with the mean difference and a 95% confidence interval for the difference. Chest wall compartments will be measured using opto-electronic plethysmography, with units in [%VT - Tidal volume], and the outcomes will be compared using a repeated-measures ANOVA with intra-subject comparisons.
Breathing frequency | up to 12 weeks
  Breathing frequency in each phase of the GXT will be presented as a mean and standard deviation, along with the mean difference and a 95% confidence interval for the difference. Breathing frequency will be measured using opto-electronic plethysmography, with units in [bpm], and the outcomes will be compared using a repeated-measures ANOVA with intra-subject comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: David Marko, Mgr, Principal Investigator — University of South Bohemia
Locations (1):
- University of South Bohemia, České Budějovice, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Au SCL. The model of N95 face mask used and hypercapnia proof upon choroidal thickness measurement. Photodiagnosis Photodyn Ther. 2021 Sep;35:102399. doi: 10.1016/j.pdpdt.2021.102399. Epub 2021 Jun 11. No abstract available. PMID 34126242
- [Background] Aliverti A, Rodger K, Dellaca RL, Stevenson N, Lo Mauro A, Pedotti A, Calverley PM. Effect of salbutamol on lung function and chest wall volumes at rest and during exercise in COPD. Thorax. 2005 Nov;60(11):916-24. doi: 10.1136/thx.2004.037937. Epub 2005 Jun 30. PMID 15994253
- [Background] Vogiatzis I, Aliverti A, Golemati S, Georgiadou O, Lomauro A, Kosmas E, Kastanakis E, Roussos C. Respiratory kinematics by optoelectronic plethysmography during exercise in men and women. Eur J Appl Physiol. 2005 Mar;93(5-6):581-7. doi: 10.1007/s00421-004-1249-4. Epub 2004 Dec 1. PMID 15578206
- [Background] Aliabadi M, Aghamiri ZS, Farhadian M, Shafiee Motlagh M, Hamidi Nahrani M. The Influence of Face Masks on Verbal Communication in Persian in the Presence of Background Noise in Healthcare Staff. Acoust Aust. 2022;50(1):127-137. doi: 10.1007/s40857-021-00260-3. Epub 2022 Jan 26. PMID 35095185
- [Background] Redlinger RE Jr, Kelly RE, Nuss D, Goretsky M, Kuhn MA, Sullivan K, Wootton AE, Ebel A, Obermeyer RJ. Regional chest wall motion dysfunction in patients with pectus excavatum demonstrated via optoelectronic plethysmography. J Pediatr Surg. 2011 Jun;46(6):1172-6. doi: 10.1016/j.jpedsurg.2011.03.047. PMID 21683217
- [Background] Wilson RC, Jones PW. A comparison of the visual analogue scale and modified Borg scale for the measurement of dyspnoea during exercise. Clin Sci (Lond). 1989 Mar;76(3):277-82. doi: 10.1042/cs0760277. PMID 2924519